CLINICAL TRIAL: NCT06946810
Title: Impact of Two TRAnsition Programs on Transition Readiness and Quality of Life in Inflammatory Bowel Disease: a Randomized Controlled Trial
Brief Title: Impact of Transition Programs on Readiness and Quality of Life in IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, ZINGONE FABIANA, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5385/AO/22
Record Dates: First submitted 2025-04-12; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Transition; Pediatric; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letter-based transition group (Active Comparator): In this arm, patients are transitioned from pediatric to adult gastroenterology care through a referral system where the pediatrician prepares a comprehensive clinical report that accompanies the patient to their first adult gastroenterology appointment. The transition occurs without joint visits between pediatric and adult specialists.
  Interventions: Behavioral: Letter-based transition
- Combined visits-based transition (Experimental): In this arm, patients experience a gradual transition involving joint consultations where both pediatric and adult gastroenterologists are present. This includes at least one combined visit at the pediatric clinic and one at the adult clinic, allowing for collaborative care and direct communication between all parties during the transition process.
  Interventions: Behavioral: Combined visits-based transition

INTERVENTIONS:
Behavioral: Combined visits-based transition — In this arm, patients experience a gradual transition involving joint consultations where both pediatric and adult gastroenterologists are present. This includes at least one combined visit at the pediatric clinic and one at the adult clinic, allowing for collaborative care and direct communication between all parties during the transition process.
  Arms: Combined visits-based transition
Behavioral: Letter-based transition — In this arm, patients are transitioned from pediatric to adult gastroenterology care through a referral system where the pediatrician prepares a comprehensive clinical report that accompanies the patient to their first adult gastroenterology appointment. The transition occurs without joint visits between pediatric and adult specialists.
  Arms: Letter-based transition group

SUMMARY:
This study is a randomized controlled trial comparing two transition models for adolescents with inflammatory bowel disease (IBD) moving from pediatric to adult care. Patients aged 16-19 years with IBD will be randomized to either a letter-based transition approach (involving a referral supported by a pediatrician's clinical report) or a combined visits-based approach (including joint consultations with both pediatric and adult gastroenterologists).

The primary outcome will be transition readiness assessed using the Transition Readiness Assessment Questionnaire (TRAQ). Secondary outcomes include quality of life (measured by the Pediatric Quality of Life Inventory™), disease activity, and healthcare utilization. Participants will be evaluated at baseline, six months, and one year. The study aims to establish an evidence-based transition model by determining which approach better facilitates a successful transition from pediatric to adult gastroenterology care for young patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* IBD diagnosis according to current guidelines
* Age between 16 and 19 years
* Disease in clinical remission or with mild activity

Exclusion Criteria:

- Subjects unable to provide a free and valid consent to study participation

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Transition readiness as measured by the Transition Readiness Assessment Questionnaire (TRAQ) | Baseline and at end of transition period (approximately 12 months)
  The TRAQ is a validated 20-item questionnaire that assesses youths' ability to manage their health independently. It evaluates five domains: Appointment Keeping, Tracking Health Issues, Managing Medications, Talking with Providers, and Managing Daily Activities. Scores range from 1-5 for each item, with higher scores indicating greater transition readiness.

SECONDARY OUTCOMES:
Quality of life as measured by the Pediatric Quality of Life Inventory™ (PedsQL™) | Baseline (Day 0), intermediate visit (Month 6), and end of transition period (Month 12)
  The PedsQL™ measures health-related quality of life in healthy children and adolescents and those with chronic conditions. It includes Physical, Emotional, Social, and School Functioning domains with scores ranging from 0-100, where higher scores indicate better quality of life.
Healthcare utilization | Throughout study period (Month 0 to Month 12)
  Tracking of hospitalizations, surgeries, and unplanned healthcare visits related to IBD during the transition period.
Quality of life as measured by the Pediatric Quality of Life Inventory™ (PedsQL™) | Baseline (T0), intermediate visit (T2), and end of transition period (T3, approximately 12 months)
  The PedsQL™ measures health-related quality of life in healthy children and adolescents and those with chronic conditions. It includes Physical, Emotional, Social, and School Functioning domains with scores ranging from 0-100, where higher scores indicate better quality of life.
Disease activity in Crohn's Disease patients | Baseline (Day 0), intermediate visit (Month 6), and end of transition period (Month 12)
  Disease activity will be measured using the Pediatric Crohn's Disease Activity Index (PCDAI) for pediatric patients or Harvey-Bradshaw Index (HBI) for adult patients. PCDAI scores range from 0-100 with remission defined as <10; HBI scores range from 0-25+ with remission defined as <5. For both scales, higher scores indicate more severe disease activity.
Disease activity in Ulcerative Colitis patients | Baseline (Day 0), intermediate visit (Month 6), and end of transition period (Month 12)
  Disease activity will be measured using the Pediatric Ulcerative Colitis Activity Index (PUCAI) for pediatric patients or partial Mayo score for adult patients. PUCAI scores range from 0-85 with remission defined as <10; partial Mayo scores range from 0-9 with remission defined as 0-1. For both scales, higher scores indicate more severe disease activity.
C-reactive protein (CRP) levels | Baseline (Day 0), intermediate visit (Month 6), and end of transition period (Month 12)
  Blood concentration of CRP measured in mg/dL as an objective marker of inflammation. Normal value is <0.5 mg/dL, with higher values indicating active inflammation.
Fecal calprotectin levels | Baseline (Day 0), intermediate visit (Month 6), and end of transition period (Month 12)
  Concentration of fecal calprotectin measured in mg/Kg as an objective marker of intestinal inflammation. Normal value is <250 mg/Kg, with higher values indicating active intestinal inflammation.
Incidence of treatment modifications | Throughout study period (Month 0 to Month 12)
  The number and type of changes in medical management (medication additions, discontinuations, or dosage adjustments) initiated during the transition period.
Transition readiness perception | Baseline (Day 0)
  Visual Analog Scale (VAS) scores from patients, parents, and pediatricians assessing perception of readiness for transition. Scores range from 0-10, with higher scores indicating greater perceived readiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale - Università Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol